CLINICAL TRIAL: NCT04150354
Title: Mental Health Symptom Monitoring Utilizing the Cogito Behavioral Analytic Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Brenner, Director of the VHA Rocky Mountain MIRECC, VA Eastern Colorado Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-0109
Record Dates: First submitted 2019-07-23; First posted 2019-11-04 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Mobile Applications; Cell Phone Use; Mental Health Issue; Acceptability of Health Care; Feasibility
MeSH Terms: conditions — Cell Phone Use; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants allocated to Cogito Companion (Experimental): Participants will have access the Cogito Companion for a three-month period post-consent. Passive data collection will also occur during this period. As a secure, privacy-compliant mobile app, the Cogito Companion facilitates the non-invasive collection, transfer, integration, analysis, and reporting of objective behavioral indicators.
  Interventions: Behavioral: Cogito Companion

INTERVENTIONS:
Behavioral: Cogito Companion — During the course of the study, the research application (Cogito Companion) will be installed on participants' mobile phone. The application on the participants' phone will be recording data about their behavior. Participants will also be asked to complete bi-weekly surveys via the app.

SUMMARY:
The primary objective of this project is to test the acceptability and feasibility of a mobile application to facilitate mental health symptom monitoring and follow-up among Veterans. During the course of the study, the research application will be installed on participants' mobile phone. The application on the participants' phone will be recording data about their behavior. Participants will also be asked to complete bi-weekly surveys via the app.

ELIGIBILITY:
Inclusion Criteria:

* Veterans between the ages 18-89 years of age at the time of enrollment
* able to provide signed and dated informed consent
* has anandroid platform phone and is willing to use phone and personal data plan to participate

Exclusion Criteria:

* Participation in conflicting Rocky Mountain MIRECC interventional protocol

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire -8 | 3 months
  Veterans' satisfaction with app
Narrative Evaluation of Intervention Interview (NEII). | 3 months
  Ease of Implementation per Veterans

CONTACTS AND LOCATIONS:
Locations (1):
- VAECHCS, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No